CLINICAL TRIAL: NCT01382862
Title: PHANTOM-S: The Pre-Hospital Acute Neurological Therapy and Optimization of Medical Care in Stroke Patients - Study
Acronym: PHANTOM-S
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Berlin Firebrigade (Unknown); MEYTEC GmbH (Unknown); B.R.A.H.M.S GmbH ThermoFisher Scientific (Unknown); Federal Ministry of Education and Research via Center for Stroke Research Berlin (CSB) (Unknown); European Union (Other); Berlin Technology Foundation (EFRE) (Unknown); The Volkswagen Foundation (Other); German Research Foundation (Other)
Responsible Party: Heinrich Audebert/ Prof. Dr. med., Charité - Universitätsmedizin Berlin, Center for Stroke Research Berlin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PHANTOM-S
Record Dates: First submitted 2011-06-21; First posted 2011-06-27 (Estimated); Last update posted 2015-09-15 (Estimated); Status verified 2013-02

CONDITIONS: Acute Stroke
Keywords: acute ischemic stroke; thrombolysis; prehospital; emergency medicine; suspected acute stroke; telemedicine
MeSH Terms: conditions — Stroke; Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Regular Care (No Intervention): Regular care for suspected stroke in Berlin consists of an ambulance with paramedics only, and neither computed tomography (CT) nor point-of-care diagnostics. In Berlin, emergency physicians are involved in prehospital care only in cases of special medical emergencies such as severe instability of vital parameters or loss of consciousness.
- Stroke Emergency Unit Mobile (STEMO) (Active Comparator): The STEMO is equipped with a CT-scanner, a point-of-care laboratory and the infrastructure for tele-radiological as well as videoconferencing support. STEMO is operated by a team of experienced neurologists (n=6, half-time positions, with additional formal training in emergency medicine according to the requirements of the Berlin Medical Board), paramedics of the fire brigade (n=3, two years formal training in emergency care) and radiology technicians (n=3, three years formal training in radiology assistance and three months formal training in emergency care).
  Interventions: Other: Stroke Emergency Mobile Unit (STEMO)

INTERVENTIONS:
Other: Stroke Emergency Mobile Unit (STEMO) — Patients treated in the STEMO may receive a CT-scan and point-of-care laboratory work up. This depends on the results of the neurological examination including assessment of medical history and the indication for scanning by the radiologist on call. In case of no contraindications patients with acute ischemic stroke will receive intravenous tissue Plasminogen Activator (0.9 mg/kg BW) according to the routine use of tissue Plasminogen Activator in Germany within 4.5 hours of symptom onset but with no formal upper age limit. (In other words, patients older than 80 years will not be excluded.) In case of increased INR and intracerebral hemorrhage patients will receive Prothrombin Complex Concentrate (PCC). All other indications will be treated according to national guidelines or as considered appropriate by the neurologist.
  Other Names: pre-hospital thrombolysis
  Arms: Stroke Emergency Unit Mobile (STEMO)

SUMMARY:
The purpose of this prospective study in acute ischemic stroke patients is to compare alarm-to-needle time during randomly allocated periods with and without availability of a specially staffed ambulance equipped with computed tomography (CT) and point-of care diagnostics. The investigators hypothesize that compared to regular care the investigators will reduce alarm-to-needle time by a minimum of 20 minutes by implementation of the stroke emergency mobile unit.

DETAILED DESCRIPTION:
Time from symptom onset is crucial for the effectiveness of intravenous thrombolysis in acute ischemic stroke patients. Many patients receive tissue Plasminogen Activator (tPA) with considerable delay. The investigators developed an ambulance equipped with a CT-scanner, point-of-care laboratory, teleradiological support and an emergency trained neurologist on board. In the Pre-Hospital Acute Neurological Therapy and Optimization of Medical care in Stroke patients (PHANTOM-S)-study the investigators aim at a reduction of the current alarm-to-needle time by pre-hospital use of tissue Plasminogen Activator in an ambulance.

The investigators hypothesize that compared to regular care we will reduce alarm-to-needle time by a minimum of 20 minutes by implementation of the stroke emergency mobile unit (STEMO).

This is a prospective study comparing randomly allocated periods with and without STEMO availability.

ELIGIBILITY:
Inclusion Criteria:

* Patients whose emergency call prompted the suspicion of stroke within 4 hours of symptom onset or with undetermined time of onset in the dispatch center
* Informed consent for documentation and follow-up provided by patients or legal representatives

Exclusion Criteria:

* age < 18 years
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 614 (Actual)
Dates: Start 2011-05; Primary Completion 2013-01 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
alarm-to-needle time | day 1
  Primary endpoint of the study is the time between activation of the emergency medical service and initiation of thrombolysis (alarm-to-needle time).

SECONDARY OUTCOMES:
Functional outcomes | three months after symptom onset
  Functional outcome of patients will be assessed via modified Rankin Scale (mRS) during telephone follow-up after three months and mortality
other times | day 1
  Alarm-to-imaging Imaging-to-needle Alarm-to-point-of-care laboratory diagnostics (International Normalized Ratio (INR), platelet count) Alarm-to-INR normalization (<1.5) in cases of intracerebral hemorrhage (ICH) and INR>1.7
Costs effectiveness will be assessed | 15 months (coinciding with the anticipated date of the completion of the last follow-up)
Proportion of stroke patients receiving tissue Plasminogen Activator (tPA) | day 1
  Proportion of stroke patients receiving tPA will be assessed and compared between regular care and STEMO.
Special referral | day 1
  Proportion of patients referred to specialized centres in case of:
  Occlusion of distal carotid / proximal middle cerebral artery Space occupying cerebellar ICH (at least 6 mL) Intraventricular haemorrhage (>/= 1 ventricle filled with blood)
symptomatic intracerebral hemorrhage | 36 hours after symptom onset
  symptomatic intracerebral hemorrhage (sICH) will be assessed according to European Cooperative Acute Stroke Study (ECASS) III and National Institute of Neurological Disorders and Stroke (NINDS) definition
Serious adverse events | up to 3 months
  Number of Serious Adverse Events (SAE) according to good clinical practice (GCP) classification
Mortality | up to three months
  In-hospital mortality (i.e. 7-days-mortality = primary safety outcome; safety analyses will include patients who received tissue Plasminogen Activator during the pilot phase of the study) and mortality three months after stroke will be assessed in stroke patients.

OTHER OUTCOMES:
Proportions of patients treated in time intervals from onset | day 1
  According to time intervals 0-90, 91-180, 181-270 minutes as used in the pooled analysis of randomized controlled iv tPA trials(K. Lees et al., Lancet, 2010).
  This outcome was specified before completion of data collection and will be used for cost-effectiveness analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Heinrich Audebert, Prof, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charite - Universitätsmedizin Berlin, Berlin, State of Berlin, Germany

REFERENCES:
- [Derived] Koch PM, Kunz A, Ebinger M, Geisler F, Rozanski M, Waldschmidt C, Weber JE, Wendt M, Winter B, Zieschang K, Bollweg K, Kaczmarek S, Endres M, Audebert HJ. Influence of Distance to Scene on Time to Thrombolysis in a Specialized Stroke Ambulance. Stroke. 2016 Aug;47(8):2136-40. doi: 10.1161/STROKEAHA.116.013057. Epub 2016 Jun 21. PMID 27328702
- [Derived] Wendt M, Ebinger M, Kunz A, Rozanski M, Waldschmidt C, Weber JE, Winter B, Koch PM, Nolte CH, Hertel S, Ziera T, Audebert HJ; STEMO Consortium. Copeptin Levels in Patients With Acute Ischemic Stroke and Stroke Mimics. Stroke. 2015 Sep;46(9):2426-31. doi: 10.1161/STROKEAHA.115.009877. Epub 2015 Aug 6. PMID 26251255
- [Derived] Wendt M, Ebinger M, Kunz A, Rozanski M, Waldschmidt C, Weber JE, Winter B, Koch PM, Freitag E, Reich J, Schremmer D, Audebert HJ; STEMO Consortium. Improved prehospital triage of patients with stroke in a specialized stroke ambulance: results of the pre-hospital acute neurological therapy and optimization of medical care in stroke study. Stroke. 2015 Mar;46(3):740-5. doi: 10.1161/STROKEAHA.114.008159. Epub 2015 Jan 29. PMID 25634000
- [Derived] Ebinger M, Kunz A, Wendt M, Rozanski M, Winter B, Waldschmidt C, Weber J, Villringer K, Fiebach JB, Audebert HJ. Effects of golden hour thrombolysis: a Prehospital Acute Neurological Treatment and Optimization of Medical Care in Stroke (PHANTOM-S) substudy. JAMA Neurol. 2015 Jan;72(1):25-30. doi: 10.1001/jamaneurol.2014.3188. PMID 25402214
- [Derived] Ebinger M, Winter B, Wendt M, Weber JE, Waldschmidt C, Rozanski M, Kunz A, Koch P, Kellner PA, Gierhake D, Villringer K, Fiebach JB, Grittner U, Hartmann A, Mackert BM, Endres M, Audebert HJ; STEMO Consortium. Effect of the use of ambulance-based thrombolysis on time to thrombolysis in acute ischemic stroke: a randomized clinical trial. JAMA. 2014 Apr 23-30;311(16):1622-31. doi: 10.1001/jama.2014.2850. PMID 24756512